CLINICAL TRIAL: NCT00851630
Title: A Pilot Study Of Open-Label Fixed Dose Combination Zidovudine/Lamivudine/Abacavir In HIV-Infected Persons With Tuberculosis In Moshi, Tanzania; Tuberculosis And HIV Immune Reconstitution Syndrome Trial (THIRST)
Brief Title: Tuberculosis and Human Immunodeficiency Virus (HIV) Immune Reconstitution Syndrome Trial (THIRST)
Acronym: THIRST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Kibongoto National Tuberculosis Hospital, Tanzania (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Nathan Thielman, MD, MPH, Duke University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013131
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2010-01-08 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: HIV; Tuberculosis
Keywords: HIV; Tuberculosis; Treatment Naive
MeSH Terms: conditions — Tuberculosis | interventions — Lamivudine; abacavir; abacavir, lamivudine, and zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early (Experimental): Initiation of fixed dose combination zidovudine/lamivudine/abacavir 2 weeks after commencing antituberculous therapy
  Interventions: Drug: Fixed dose combination zidovudine/lamivudine/abacavir
- Delayed (Experimental): Initiation of fixed dose combination zidovudine/lamivudine/abacavir 8 weeks after commencing antituberculous therapy
  Interventions: Drug: Fixed dose combination zidovudine/lamivudine/abacavir

INTERVENTIONS:
Drug: Fixed dose combination zidovudine/lamivudine/abacavir — All subjects will receive fixed dose combination zidovudine(300 mg) / lamivudine (150 mg) / abacavir (300 mg) by mouth twice daily. Medications will be provided as long as deemed beneficial by the site investigator and study subject for up to two years. Toxicity substitutions are allowed per protocol.
  Other Names: Trizivir

SUMMARY:
The purpose of this study is twofold: (1) to assess the feasibility and safety of fixed dose combination zidovudine/lamivudine/abacavir in HIV infected subjects with tuberculosis in a resource-limited setting, and (2) to assess the impact of delayed versus early initiation strategies for fixed dose combination zidovudine/lamivudine/abacavir on the rate of tuberculosis-associated immune reconstitution inflammatory syndromes.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infection is documented by rapid HIV test or any licensed enzyme-linked immunosorbent assay (ELISA) test kit and confirmed with a different sample.
* Men or women admitted to Kibongoto or Marangu Hospitals with (a) recent (within 56 days) smear positive tuberculosis (pulmonary or extrapulmonary,) (b)total lymphocyte count <1,200/mm3, and (c) less than 14 days of antituberculous therapy.
* Antiretroviral naive with the exception of regimens used to prevent mother-to-infant transmission of HIV during pregnancy.
* The following laboratory values obtained within 45 days prior to study entry: absolute neutrophil count (ANC) >=700/mm³, hemoglobin > 8 g/dL in women; >9 g/dL in men, serum creatinine <= 1.5 times upper limits of normal, AST <5 times upper limits of normal.
* For all women of reproductive potential (who have not reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation), a negative urine pregnancy test within 48 hours of to study.
* All subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate) and if participating in sexual activity that could lead to pregnancy, the female subject/male partner must use condoms (male or female) without a spermicidal agent.
* Not intending to relocate out of area for the duration of study participation.
* Willingness of subject to adhere to follow up schedule.
* Men and women >= age 13.
* Ability and willingness of subject or legal guardian/representative to give written consent.

Exclusion Criteria:

* Serious illness, other than tuberculosis, that requires systematic treatment and/or hospitalization, until either completion of therapy or clinical stability on therapy in the opinion of the investigator for at least 14 days prior to study entry. Oral and vaginal candidiasis, mucocutaneous herpes simples, and other illnesses which are minor in the opinion of the site investigator are exceptions
* Diagnosis of or suspicion of tuberculosis of the central nervous system.
* > 14 days of antituberculous therapy prior to screening.
* > 28 days of antituberculous therapy for active tuberculosis within the 6 months prior to screening.
* Recent past (within 28 days of study entry) or planned use of corticosteroids.
* Any condition that in the opinion of the investigator would compromise the subject's ability to participate in the study.
* Radiation or systemic chemotherapy within 45 days of entry.
* Any immunomodulator, HIV vaccine, or other investigational therapy within 30 days prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Allergy/sensitivity to any study drugs or their formulations.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan M Thielman, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

REFERENCES:
- [Result] Shao HJ, Crump JA, Ramadhani HO, Uiso LO, Ole-Nguyaine S, Moon AM, Kiwera RA, Woods CW, Shao JF, Bartlett JA, Thielman NM. Early versus delayed fixed dose combination abacavir/lamivudine/zidovudine in patients with HIV and tuberculosis in Tanzania. AIDS Res Hum Retroviruses. 2009 Dec;25(12):1277-85. doi: 10.1089/aid.2009.0100. PMID 20001518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in June 2004 and was completed in September 2005. Patients were enrolled at one of two hospitals in the Kilimanjaro Region of Tanzania.
Groups:
- Early: Initiation of fixed dose combination zidovudine (300 mg)/lamivudine (150 mg)/abacavir (300 mg) administered orally twice daily, beginning 2 weeks after commencing antituberculous therapy
- Delayed: Initiation of fixed dose combination zidovudine (300 mg)/lamivudine (150 mg)/abacavir (300 mg) administered orally twice daily, beginning 8 weeks after commencing antituberculous therapy
Period: Overall Study
Arm/Group | Early | Delayed
Started | 35 | 35
Completed | 33 | 33
Not Completed | 2 | 2
Not completed — Death | 2 | 1
Not completed — Clinical failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early | Delayed | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1.0
  Between 18 and 65 years | 34 | 35 | 69.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Median (Inter-Quartile Range); unit: years] | 36.0 [32.4 to 43.6] | 36.7 [32.4 to 44.3] | 36.2 [32.4 to 43.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29.0
  Male | 23 | 18 | 41.0
Region of Enrollment [Number; unit: participants]
  Tanzania | 35 | 35 | 70.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events (SAEs)
Description: Feasibility and safety of fixed dose combination zidovudine/lamivudine/abacavir in HIV-infected subjects with tuberculosis in a resource-limited setting as assessed by the number of serious adverse events. Serious adverse events included any untoward medical occurrence that resulted in death, was considered life-threatening, required inpatient hospitalization or prolongation of existing hospitalization beyond what was required in the study, or resulted in persistent or resulted in significant disability/incapacity.
Time Frame: 104 weeks
Population: Intention to treat.
Measure: Number; unit: Events
Arm/Group | Early | Delayed
Number analyzed (Participants) | 35 | 35
Events | 12 | 7

2. Primary Outcome: Tuberculosis-immune Reconstitution Inflammatory Syndrome Events
Description: Tuberculosis-immune reconstitution inflammatory syndrome was defined by the protocol as: a) new persistent fevers (temperature >101.5 degrees Fahrenheit) developing after the initiation of antiretroviral therapy, and not believed to be associated with antiretroviral therapy and without an identifiable source, b) marked worsening or emergence of intrathoracic lymphadenopathy, pulmonary infiltrates or pleural effusions on radiologic examination, or c) worsening or emergence of lymphadenopathy on serial examinations or worsening of other tuberculous lesions.
Time Frame: 104 weeks
Population: Intention to treat.
Measure: Number; unit: Events
Arm/Group | Early | Delayed
Number analyzed (Participants) | 35 | 35
Events | 0 | 0

3. Secondary Outcome: Plasma HIV Ribonucleic Acid (RNA) Level < 400 Copies/ml
Description: The number of subjects with plasma HIV RNA level <400 copies/ml.
Time Frame: 104 Weeks
Population: Intention to Treat Analysis, missing = failure.
Measure: Number; unit: Participants
Arm/Group | Early | Delayed
Number analyzed (Participants) | 35 | 35
Participants | 26 | 31

4. Secondary Outcome: HIV RNA Level < 50 Copies/ml
Description: The number of subjects with plasma HIV RNA level <50 copies/ml.
Time Frame: 104 Weeks
Population: Intent to Treat, missing = failure.
Measure: Number; unit: Participants
Arm/Group | Early | Delayed
Number analyzed (Participants) | 35 | 35
Participants | 23 | 26

ADVERSE EVENTS:
Arm/Group | Early | Delayed
Serious Adverse Events (participants affected / at risk) | 12/35 | 7/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early (N=35) | Delayed (N=35)
Acute intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Allergic reaction to suphalene-pyrimethamine (Immune system disorders) | 0 (0) | 1 (1)
Amebiasis (Infections and infestations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cryptococcal meningitis (Infections and infestations) | 1 (1) | 0 (0)
Disseminated kaposi's sarcoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Esophageal variceal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Head trauma, grand mal seizure (Nervous system disorders) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 2 (2) | 1 (1)
Mycobacteremia with M. sherrisii (Infections and infestations) | 0 (0) | 1 (1)
Suspected abacavir hypersensitivity reaction (Immune system disorders) | 3 (3) | 1 (1)
Syphilis (Infections and infestations) | 1 (1) | 0 (0)
Tension pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No